CLINICAL TRIAL: NCT00897741
Title: Gene Expression Profiles in Primary and Metastatic Pancreatic Cancer
Brief Title: Gene Expression Profiles in Patients With Metastatic Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000482353; P30CA022453 (NIH); WSU-D-2841; WSU-HIC-091504M1E
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study uses gene expression profiling to compare primary tumor cells with metastatic tumor cells in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the gene expression profiles of pancreatic cancer cells from the primary and metastatic sites in patients with metastatic pancreatic cancer.
* Characterize the function of the differentially upregulated and downregulated genes identified by comparing the gene expression profiles of primary and metastatic cells in these patients.

OUTLINE: Fresh biopsy samples are collected for gene expression profiling and other biomarker/laboratory analyses.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pancreatic adenocarcinoma of exocrine origin
* Metastatic disease
* Fresh biopsy material available from primary site of disease and a metastatic focus, including liver, peritoneum, or lymph node

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for pancreatic cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Gene expression profiles | at time of biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States